CLINICAL TRIAL: NCT05489887
Title: A Phase II Study of Naxitamab Added to Induction Therapy for Subjects With Newly Diagnosed High-Risk Neuroblastoma
Brief Title: Naxitamab Added to Induction for Newly Diagnosed High-Risk Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC018
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma
Keywords: naxitimab; induction
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HRNB Newly diagnosed subjects (Experimental): 5 cycles of standard of care induction + naxitimab
  Naxitimab on Days 1, 3, and 5 of each cycle
  Interventions: Drug: Naxitamab

INTERVENTIONS:
Drug: Naxitamab — Naxitamab is a humanized (IgG1) anti-GD2 (hu3F8) monoclonal antibody for the treatment of neuroblastoma, osteosarcoma and other GD2-positive cancers. Naxitamab was granted accelerated approval by the FDA in 2020 as treatment (in combination with granulocyte-macrophage colony-stimulating factor - GM-CSF) for pediatric patients at least one year of age and adult patients with relapsed or refractory high-risk neuroblastoma in the bone or bone marrow demonstrating a partial response, minor response, or stable disease to prior therapy
  Other Names: Danyelza

SUMMARY:
This is a prospective, multicenter clinical trial in subjects with newly diagnosed high-risk neuroblastoma to evaluate the efficacy and safety of administering naxitamab with standard induction therapy. The initial chemotherapy will include 5 cycles of multi-agent chemotherapy. Naxitamab will be added to all 5 Induction cycles. We hypothesize that the addition of anti-GD2 therapy to induction chemotherapy will result in improved end of induction responses and improved survival.

DETAILED DESCRIPTION:
This is a prospective, multicenter clinical trial in subjects with newly diagnosed high-risk neuroblastoma to evaluate the efficacy and safety of administering naxitamab with standard induction therapy.

All subjects will be followed for disease response, event free survival, overall survival and toxicity. Extent of disease will be measured and assessed for changes throughout the course of the study. All efficacy analyses will be performed on the evaluable population which will consist of all enrolled subjects (subjects who initiate treatment with naxitamab in combination with GM-CSF plus standard induction therapy) and who have measurable disease at baseline.

The initial chemotherapy Induction regimen will utilize sequential administration of 5 cycles of multi-agent chemotherapy. Naxitamab will be added to all 5 Induction cycles.

Stem cell mobilization and collection will occur after the 2nd cycle of induction.

Surgical resection of the primary tumor will ideally occur after the 4th cycle of Induction but may be delayed until after the 5th cycle of Induction if medically necessary.

Disease status evaluations will occur at the following time points: (1) pre-treatment, (2) post Cycle 2 Induction (3) Prior to surgical resection (if performed), (4) End of Induction (which includes surgery and 5 cycles of chemotherapy), and (5) End of Additional/Salvage Therapy as needed.

The current standard of care for high-risk neuroblastoma involves 5-7 cycles of induction chemotherapy with surgical removal of the tumor after 4-5 cycles of chemotherapy, followed by high-dose chemotherapy plus autologous stem cell transplant, then radiation to the primary tumor bed, followed by anti-GD2 immunotherapy and cis retinoic acid. This results in a less than 60% disease free survival for high-risk NB, a survival rate that still greatly needs improvement. Two areas in which improvements can be made include: 1) to improve response rate to induction chemotherapy and 2) to improve EFS by improving maintenance therapy to prevent relapse.

We hypothesize that the addition of anti-GD2 therapy to induction chemotherapy will result in improved end of induction responses and improved survival.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Subjects must have a diagnosis of neuroblastoma or ganglioneuroblastoma (nodular or intermixed) verified by histology or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites. Subjects with the following disease stages at diagnosis are eligible, if they meet the other specified criteria:
2. Subjects with newly diagnosed neuroblastoma with INRGSS Stage M disease with either of the following features:

   1. MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of additional biologic features; OR
   2. 365 days to ≥ 547 days of age without MYCN amplification, but unfavorable biologic features such as unfavorable histology (INPC) or diploid tumor (DNA index=1) or the presence of any segmental chromosome aberration (SCA) (somatic copy number loss at 1p, 3p, 4p, or 11q or somatic copy number gain at 1q, 2p, or 17q); OR
   3. Age > 547 days of age regardless of biologic features

   Subjects with newly diagnosed neuroblastoma with INRGSS Stage MS disease with either of the following:
   1. MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals); OR
   2. 365 days to ≥ 547 days (18 months) of age without MYCN amplification, but unfavorable biologic features such as unfavorable histology (INPC) or diploid tumor (DNA index=1) or SCA as above

   Subjects with newly diagnosed neuroblastoma INRGSS Stage L2 disease with either of the following:
   1. MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals); OR
   2. 18 months to <5 years of age without MYCN amplification, but with unfavorable histology (INPC); OR
   3. ≥5 years of age without MYCN amplification, but with undifferentiated or poorly differentiated INPC Subjects with newly diagnosed neuroblastoma INRGSS Stage L1 disease that is incompletely resected with MYCN amplification.

   Subjects > 547 days of age initially diagnosed with INRGSS Stage L1, L2 or MS disease who progressed to Stage M without prior chemotherapy may enroll within 4 weeks of progression to Stage M.

   Subjects ≥ 365 days of age initially diagnosed with MYCN amplified INRGSS Stage L1 disease who progress to Stage M without systemic therapy may enroll within 4 weeks of progression to Stage M.
3. Subjects must be age ≤ 21 years at initial diagnosis.
4. Subjects must be >12 months of age at enrollment.
5. Adequate cardiac function defined as:

   1. Shortening fraction of ≥ 27% by echocardiogram, or
   2. Ejection fraction of ≥ 50% by radionuclide evaluation or echocardiogram.
6. Adequate liver function must be demonstrated, defined as:

   1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND
   2. ALT (SGPT) < 5 x upper limit of normal (ULN) for age
7. Subjects must have adequate renal function defined as an estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70.

   The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr
8. A negative serum pregnancy test is required for female participants of childbearing potential (≥13 years of age or after onset of menses)
9. Both male and female post-pubertal study subjects must be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) from the time of informed consent until 6 months after study treatment discontinuation. Such methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence.
10. Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Subjects who are less than 1 year of age
2. Subjects who are 12-18 months of age with INRGSS Stage M and all stage L2 subjects with favorable biologic features (i.e., nonamplified MYCN, favorable pathology, and DNA index > 1) are not eligible.
3. Subjects who have had prior systemic therapy except for localized emergency radiation to sites of life-threatening or function-threatening disease and/or no more than 1 cycle of chemotherapy.
4. Treatment with immunosuppressive treatment (topical, inhaled and short-term emergency steroids excluded) within 4 weeks prior to enrollment
5. Inadequate pulmonary function defined as evidence of dyspnea at rest, exercise intolerance, and/or chronic oxygen requirement. In addition, room air pulse oximetry < 94% and/or abnormal pulmonary function tests if these assessments are clinically indicated.
6. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study.)
7. Subjects receiving any investigational drug concurrently.
8. Subjects with any other medical condition, including but not limited to malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a subject's ability to sign or the legal guardian's ability to sign the informed consent, and subject's ability to cooperate and participate in the study
9. Subjects with a significant intercurrent illness (any ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and that is expected to interfere with the action of investigational medicinal products (IMPs) or to significantly increase the severity of the toxicities experienced from trial treatment.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2036-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Complete Response (CR) rate per 1993 INRC guidelines | 6 to 12 months
  Measured by the presence of radiologically assessable disease by cross-sectional computed tomography (CT) or Magnetic resonance imaging (MRI) imaging and/or by metaiodobenzylguanidine (MIBG) or positron emission tomography (PET) scans and bone marrow (BM) response for subjects with newly-diagnosed high-risk neuroblastoma according to the 1993 International Neuroblastoma Response Criteria (INRC) and compare to relevant historical controls.

SECONDARY OUTCOMES:
Number of participants with CR + Very Good Partial Response (VGPR) rate and objective response rate (ORR; CR + VGPR + PR) | 6 to 12 months
  Evaluate the combined CR + Very Good Partial Response (VGPR) rate and objective response rate (ORR; CR + VGPR + PR) at EOI per 1993 INRC, compared against historical controls and external controls. Measured by the presence of radiologically assessable disease by cross-sectional computed tomography (CT) or Magnetic resonance imaging (MRI) imaging and/or by metaiodobenzylguanidine (MIBG) or positron emission tomography (PET) scans and bone marrow (BM) response for subjects with newly-diagnosed high-risk neuroblastoma according to the 1993 International Neuroblastoma Response Criteria (INRC).
Number of participants with Complete Response (CR) rate per 2017 INRC guidelines | 6 to 12 months
  Evaluate CR rate and ORR (CR + PR) at EOI per the 2017 INRC, compared against external controls. Measured by the presence of radiologically assessable disease by cross-sectional computed tomography (CT) or Magnetic resonance imaging (MRI) imaging and/or by metaiodobenzylguanidine (MIBG) or positron emission tomography (PET) scans and bone marrow (BM) response for subjects with newly-diagnosed high-risk neuroblastoma according to the 2017 International Neuroblastoma Response Criteria (INRC).
Number of days that subjects remain alive | Through study completion, an average of 1 year, plus 8 years of follow up
  Overall survival (OS) for subjects receiving the combination of standard Induction chemotherapy with naxitamab.
Number of days that subjects remain in remission | Through study completion, an average of 1 year, plus 8 years of follow up
  Progression-free survival (PFS) for subjects receiving the combination of standard Induction chemotherapy with naxitamab.
Number of participants with treatment-related adverse events | At last dose of Naxitamab, average of 6-12 months, plus 42 additional days

CONTACTS AND LOCATIONS:
Overall Officials: Jaqueline Kraveka, DO, Study Chair — Medical University of South Carolina
Locations (23):
- United States (20):
  - University of Alabama/Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Augusta University Health, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Norton Children's Research Institute/Affiliated with University of Louisville School of Medicine, Louisville, Kentucky
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (3):
  - UHC Sainte-Justine, Montreal, Quebec
  - CHUQ, Québec, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — https://research.beatcc.org/